CLINICAL TRIAL: NCT05424497
Title: Outcome, Hindsight and Implicit Bias in Emergency Medicine and Medical Disciplinary Law.
Acronym: OHIBEM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Maxima Medical Center (Other)
Responsible Party: Principal Investigator, Bart Candel, Principal Investigator, Maxima Medical Center
Other Study IDs: N22.025
Record Dates: First submitted 2022-06-07; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Emergencies; Implicit Bias
MeSH Terms: conditions — Emergencies; Bias, Implicit

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- No outcome provided
  Interventions: Other: Vignettes
- outcome positive
  Interventions: Other: Vignettes
- outcome negative
  Interventions: Other: Vignettes
- implicit bias group
  Interventions: Other: Vignettes

INTERVENTIONS:
Other: Vignettes — Presenting vignettes with fictive cases

SUMMARY:
Background Hindsight bias and outcome bias may play an important role in retrospective law of errors in Emergency Medicine and may affect judgement. In addition, differences in sex and medical history may affect treatment decisions (implicit bias).

Aims First, to assess if and to what extent knowledge of an outcome may affect the ability of Emergency Physicians and physicians with experience in disciplinary law to determine the quality of care given. Secondly, to investigate whether a medical history with nonspecific/functional/somatoform complaints and sex differences affect clinical decision making in Emergency Physicians.

Study design and analyses A web-based cross-sectional survey using vignettes with six clinical scenarios (four vignettes for outcome/hindsight bias, four vignettes for implicit bias). The survey was sent to all Emergency Physicians and residents in training in the Netherlands. Four scenarios were also sent to physicians with experience in disciplinary law. In four vignettes, participants received a scenario without an outcome, or with a positive or negative outcome. They were asked to rate the quality of care provided as sufficient or insufficient and, in more detail, poor/below average/average/good/outstanding and how likely they thought it would be that the patient would have had a negative outcome (in percent). In the other two vignettes, participants received one vignette describing a scenario of a patient presenting to the ED with acute abdominal pain and one vignette describing a scenario with chest pain. The sex and medical history differed among the participants (e.g. male/female, nonspecific medical history/somatic medical history). Participants were asked whether they would prescribe pain medication, and whether they would do diagnostic imaging.

Importance and impact This research may help to understand the impact of knowing the outcome in retrospective laws in Dutch Emergency Physicians and physicians with experience in disciplinary law. If outcome and hindsight bias are present, retrospective judgement may need a different approach in medicine, i.e. blinding judges for the outcome, to prevent wrong justice and adverse effect on clinicians well-being. Also, if implicit bias in sex and medical history is present, a training programme is needed to reduce certain bias and to improve equality in the provided care.

ELIGIBILITY:
Inclusion Criteria:

* Emergency physicians or residents, General practitioners, and physicians with experience in disciplinary law.

Exclusion Criteria:

* others

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — differences in sex in judgement and vignettes
Study Population: Emergency physicians selected through email plus physicians with experience in disciplinary law.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-06-16 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of care | Throughout the study, 1day
  The quality of care rated on a likert scale from 1 to 5 will be assessed for 4 fictive cases. The mean will be compared for each case without outcome, with positive outcome, and with negative outcome.
Diagnostic imaging | Throughout the study, 1day
  Whether the physician would perform diagnostic imaging after reading the vignette. The The outcome will be compared for vignettes including a somatic medical history with the vignettes with a nonsomatic medical history.

SECONDARY OUTCOMES:
Hindsight bias | Throughout the study, 1day
  The estimate of the chance of getting the negative outcome (0 to 100%). Compared between the group of vignettes without outcome, with a positive outcome and with a negative outcome.
Pain medication | Throughout the study, 1day
  Whether pain medication is prescribed (y/n) and how many milligrams. Compared between group of patients with somatic medical history and nonsomatic medical history.

IPD SHARING:
Plan to Share IPD: No
on request